CLINICAL TRIAL: NCT02604043
Title: Continuous Supraglottic pH Monitoring in Prolonged Intubated Intensive Care Patients and High Risk Aspiration Intraoperative Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of support to complete
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Bret Alvis, Assistant Professor Anesthesiology Critical Care Medicine, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 131893
Record Dates: First submitted 2015-11-11; First posted 2015-11-13 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Aspiration, Respiratory
Keywords: supraglottic pH
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- supraglottic impendence/pH probe (Experimental)
  Interventions: Other: pH monitoring; Other: accelerometer monitoring

INTERVENTIONS:
Other: pH monitoring — After endotracheal intubation, the impedence/pH probe will be placed under indirect visualization using a McGrath MAC video laryngoscope directly above the vocal cords. The sensor will remain in place for the duration of the surgery or for 24 hours in ICU patients. At that time, the device will be manually removed by a member of the study staff.
Other: accelerometer monitoring — Patient position will be continuously monitored with the accelerometer for the duration of the pH monitoring period.

SUMMARY:
This is a pilot prospective cohort study of the incidence of supraglottic pH readings.

DETAILED DESCRIPTION:
Aspiration is a serious morbidity that leads to an increase in both patient mortality and duration of hospital stays. Many practices exist within the hospital setting whose goal is to help prevent clinically significant aspiration including preoperative starvation, pharmaceutically reducing gastric acidity, facilitating gastric drainage, postural changes, cricoid pressure, endotracheal cuff pressure modification, and maintenance of a competent lower esophageal sphincter. However, to date, no monitoring system exists to help a clinician identify active aspiration. At present, video fluoroscopy, is the gold standard for detecting aspiration. This pilot prospective cohort study will examine the incidence of supraglottic pH readings.

A continuous pH/impedence sensor will be placed immediately above the glottic opening in four high risk populations: burn patients who are intubated, intubated post-stroke patients, patients undergoing robotic prostectomy, and in patients undergoing peritoneal tumor debulking and chemotherapy. The presence of acidic fluid above the glottic opening will be measured using a supraglottic impendence/pH probe attached to an endotracheal tube.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to undergo robotic prostatectomy.
* Patients undergoing peritoneal tumor debulking and chemotherapy
* Mechanically ventilated Burn Intensive Care Unit (BICU) Patients
* Mechanically ventilated Neuro Care Unit (NCU) Patients who have suffered a stroke

Exclusion Criteria:

* ICU patients who are not receiving enteral feeds
* Patients who present for tumor debulking or robotic prostatectomy who receive preoperative H2 blockers, proton pump inhibitors, antacids or metoclopramide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-08; Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Number of times pH drops below 5.5. | 24 hours period after placement of pH probe

SECONDARY OUTCOMES:
The mean of the angle (degrees) of the patient from the lateral position during low pH periods | 24 hours period after placement of pH probe

OTHER OUTCOMES:
Number of minutes the pH is less than 5.5 in a 24 hour | 24 hours period after placement of pH probe

CONTACTS AND LOCATIONS:
Overall Officials: Brett Alvis, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Ng A, Smith G. Gastroesophageal reflux and aspiration of gastric contents in anesthetic practice. Anesth Analg. 2001 Aug;93(2):494-513. doi: 10.1097/00000539-200108000-00050. PMID 11473886
- [Background] Clayton J, Jack CI, Ryall C, Tran J, Hilal E, Gosney M. Tracheal pH monitoring and aspiration in acute stroke. Age Ageing. 2006 Jan;35(1):47-53. doi: 10.1093/ageing/afj007. PMID 16364934